CLINICAL TRIAL: NCT03925272
Title: Constitution d'Une Cohorte Prospective de Sujets Sains et Malades et d'Une Collection de Ressources Biologiques associées Pour l'étude du système Immunitaire et de Ses déterminants Génétiques et Environnementaux"
Brief Title: Creation of a Prospective Cohort of Healthy and Sick Subjects and of a Collection of Associated Biological Resources, for the Study of the Immune System and of Its Genetic and Environmental Determinants.
Acronym: CoSImmGEn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 2010-06; 1006 (Other: Institut Pasteur)
Record Dates: First submitted 2019-04-09; First posted 2019-04-24 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Immune System and Related Disorders
Keywords: immune system; environmental interactions; genetic component
MeSH Terms: interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Who Masked: Participant

ARMS (7):
- Patients with Suppurated Hidradenitis (Experimental): Human biological samples :
  Whole blood and derived products (DNA, RNA), urine, stool, saliva, tears, skin and mouth swabs, lesion samples: swab for microbiological analyzes, cutaneous biopsies (lesion skin and peri-lesional healthy skin), surgical lesion excisions, nasal swab, oro-pharyngeal swab, nasopharyngeal swab.
  bio-clinical data: Ethno-geographical, family and personal antecedents and current events in particular related to Verneuil's disease and any associated diseases (chronic auto-inflammatory ...)
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis; Procedure: Sample obtained after surgery performed in the context of care
- Patients with Alzheimer disease (Experimental): Human biological samples :
  stool, blood (20 ml), nasal swab, oro-pharyngeal swab, nasopharyngeal swab.
  bio-clinical data: healthy or sick status,cognitive, memory and psychometric abilities evaluated by different tests example: MMSE (for Alzheimer's) and MST (minor memory disorders), Psychometric abilities assessed by the Geriatric Depression Scale GDS, Nutritional status assessed by the MNA test
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis
- Patients with familial adenomatous polyposis (Experimental): Human biological samples :
  whole blood (30 to 100 mL), optional stool collection
  bio-clinical data: Age, Gender, Ethnicity, Personal and Family Medical History, Current Treatment, Type of PAF Mutation
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis
- Patients with chronic inflammatory diseases (SPA, Crohn, ...) (Experimental): Human biological samples :
  whole blood and derived products (DNA, RNA, PBMC, plasma, serum), (100 mL), stool; as part of the treatment, occasionally: lesions, urine, saliva, tears
  Bio-clinical data :
  Ethno-geographical origin, Personal and family history, History of the disease, Associated or concomitant diseases, Treatments in progress.
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis; Procedure: Sample obtained after surgery performed in the context of care
- Healthy cases (Experimental): Human biological samples :
  whole blood and derived products: serum, plasma, DNA, RNA, PBMCs, T and B lymphocytes, monocytes / dendritic cells derived, other subpopulations (PMN, NK, etc.), urine, stool, saliva, tears, oral swabs, cutaneous swabs (healthy and injured), cutaneous biopsies (healthy and injured) and their derivatives (RNA, histological blocks ...), surgical excisions, nasal swab, oro-pharyngeal swab, nasopharyngeal swab.
  Bio-clinical data :
  ethno-geographical origin (5 groups), family and personal antecedents and contemporary events visits, in particular related to the immune system, infections, vaccinations, exposure factors (travel, lifestyles, stress, pollution cancers, allergies , chronic inflammatory diseases ...
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis
- Healthy cases relatives (Experimental): Human biological samples :
  whole blood and derived products: serum, plasma, DNA, RNA, PBMCs, T and B lymphocytes, monocytes / dendritic cells derived, other subpopulations (PMN, NK, etc.), urine, stool, saliva, tears, oral swabs, cutaneous swabs (healthy and injured), cutaneous biopsies (healthy and injured) and their derivatives (RNA, histological blocks ...), surgical excisions, nasal swab, oro-pharyngeal swab, nasopharyngeal swab.
  Bio-clinical data :
  ethno-geographical origin (5 groups), family and personal antecedents and contemporary events visits, in particular related to the immune system, infections, vaccinations, exposure factors (travel, lifestyles, stress, pollution cancers, allergies , chronic inflammatory diseases ...
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis
- Subjects vaccinated against COVID-19 (Experimental): Human biological samples :
  whole blood and derived products: serum, DNA, PBMCs, saliva, nasopharyngeal swab
  Bio-clinical data :
  ethno-geographical origin, family and personal antecedents and contemporary events visits, in particular related to the immune system, infections, vaccinations, exposure factors (travel, lifestyles, stress, pollution cancers, allergies , chronic inflammatory diseases, specific history of otorhinolaryngology and broncho-pulmonary and treatments, specific COVID-19 history, risk factor for a severe form of COVID-19, symptoms of COVID-19 or positive test for SarsCov-2 positive
  Interventions: Procedure: Collection of samples (blood, stool, etc.); Genetic: Genetic determinants analysis

INTERVENTIONS:
Procedure: Collection of samples (blood, stool, etc.)
Genetic: Genetic determinants analysis
Procedure: Sample obtained after surgery performed in the context of care
  Arms: Patients with Suppurated Hidradenitis; Patients with chronic inflammatory diseases (SPA, Crohn, ...)

SUMMARY:
CoSImmGEn is a protocol set up to respond to the current lack of healthy and sick population cohorts. Biological resources from these cohorts allow researchers to study the immune system and its genetic and environmental determinants. Those cohorts and collections are open not only to the Pasteurian community but also to the worldwide scientific community (both public and private) working in the field.

DETAILED DESCRIPTION:
The CoSImmGEn protocol is dedicated to the study of the immune system in healthy people or people with specific pathologies. It is composed of 6 arms (sub-cohorts):

* Arm "main cohort CoSImmGEn": comprised of 5 sub groups (A, B, C, D, M) of healthy adult subjects from various ethno-geographical origins.
* Arm "ancillary cohort P" comprised of first-degree relatives (including parents, siblings, or children), whether they are healthy or ill. It will allow, whenever necessary, to remove allelic ambiguities for example for the study of HLA and MHC genes.
* Arm "ancillary cohort HS": comprised of subjects suffering from Suppurativa Hidradenitis (or Verneuil's disease.) The investigators will include patients suffering from this disease and their close relatives, in order to understand the genetic, immunological, microbiological and metabolomic bases of this disease.
* Arm "ancillary cohort J": comprised of elderly patients (≥ 65 years old) with Alzheimer's disease and with mild, moderate or severe cognitive impairment. It will help understand the role of the gut microbiota in age-related brain deficits.
* Arm "ancillary cohort F": comprised of patients with familial adenomatous polyposis and carrying a mutation of the APC (Adenomatous Polyposis Coli) tumor suppressor gene. That arm has been set up to carry out a pilot phase on the role of APC mutations on anti-tumoral immune response.
* Arm "ancillary cohort I": comprised of patients with chronic inflammatory diseases such as Ankylosing spondylitis and Crohn's disease.
* Arm "ancillary cohort V": comprised of subjects vaccinated against COVID-19. It will help to follow-up the immune response after vaccination against COVID-19 in the general population.

Additional arms may be set up through new collaborations in the next few years to study others diseases in which the immune system intervenes, such as: infectious diseases, allergies or cancers.

ELIGIBILITY:
Inclusion Criteria:

* unprotected adults with social security who have attested their consent after receiving any relevant information about the study
* subjects whose ethno-geographical origin of both parents is known
* subjects for whom data on principal vaccinations (diphtheria, tetanus, poliomyelitis, hepatitis B, possibly tuberculosis) are documented
* subjects who consented to carry out serological tests HIV, HCV, HBV

Exclusion Criteria:

* Any conditions that would not allow participation in the present study, on the opinion of the investigator (documenting), ie any acute or chronic pathology that may interfere with the immune system, such as progressive or chronic pathology severe or uncontrolled by current treatments or a pathology requiring the administration of immune impact drugs: long-term anti-inflammatory, immunosuppressive, etc
* Pregnant or lactating women
* For the realization of skin biopsies: allergy to local anesthetics, cardiac valvulopathy
* For the realization of Tubertest: Subject presenting a contraindication to tuberculin

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2011-02-02 (Actual); Primary Completion 2023-12-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Immunological analysis | through study completion, an average of 4 year
  Percentage of blood cells harbouring morphological of functional abnormalities identified by flow cytometry and TrueCulture system analysis.

SECONDARY OUTCOMES:
Genetic analysis | through study completion, an average of 4 year
  Identification of genetic factors implicated in or predisposing to specific diseases through gene expression quantification, targeted genotyping of exome sequencing or whole genome sequencing.
Microbiota analysis | through study completion, an average of 4 year
  Identification of specific compositions of intestinal and/or cutaneous microbiota associated with specific diseases by metagenomic analysis.
Metabolomic analysis | through study completion, an average of 4 year
  Quantification of blood metabolites by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noelle Ungeheuer, PhD, Principal Investigator — Institut Pasteur - ICAReB
Locations (4):
- France (4):
  - Centre médical de l'Institut Pasteur, Paris
  - Institut Pasteur, Paris
  - Hopital sainte Périne, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iglesias MC, Briceno O, Gostick E, Moris A, Meaudre C, Price DA, Ungeheuer MN, Saez-Cirion A, Mallone R, Appay V. Immunodominance of HLA-B27-restricted HIV KK10-specific CD8(+) T-cells is not related to naive precursor frequency. Immunol Lett. 2013 Jan;149(1-2):119-22. doi: 10.1016/j.imlet.2012.10.002. Epub 2012 Oct 13. PMID 23068784
- [Background] Duffy D, Rouilly V, Libri V, Hasan M, Beitz B, David M, Urrutia A, Bisiaux A, Labrie ST, Dubois A, Boneca IG, Delval C, Thomas S, Rogge L, Schmolz M, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Functional analysis via standardized whole-blood stimulation systems defines the boundaries of a healthy immune response to complex stimuli. Immunity. 2014 Mar 20;40(3):436-50. doi: 10.1016/j.immuni.2014.03.002. PMID 24656047
- [Background] Thomas S, Rouilly V, Patin E, Alanio C, Dubois A, Delval C, Marquier LG, Fauchoux N, Sayegrih S, Vray M, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. The Milieu Interieur study - an integrative approach for study of human immunological variance. Clin Immunol. 2015 Apr;157(2):277-93. doi: 10.1016/j.clim.2014.12.004. Epub 2015 Jan 3. PMID 25562703
- [Background] Monceaux V, Chiche-Lapierre C, Chaput C, Witko-Sarsat V, Prevost MC, Taylor CT, Ungeheuer MN, Sansonetti PJ, Marteyn BS. Anoxia and glucose supplementation preserve neutrophil viability and function. Blood. 2016 Aug 18;128(7):993-1002. doi: 10.1182/blood-2015-11-680918. Epub 2016 Jul 8. PMID 27402974
- [Background] Urrutia A, Duffy D, Rouilly V, Posseme C, Djebali R, Illanes G, Libri V, Albaud B, Gentien D, Piasecka B, Hasan M, Fontes M, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Standardized Whole-Blood Transcriptional Profiling Enables the Deconvolution of Complex Induced Immune Responses. Cell Rep. 2016 Sep 6;16(10):2777-2791. doi: 10.1016/j.celrep.2016.08.011. Epub 2016 Aug 25. PMID 27568558
- [Background] Hamimi C, David A, Versmisse P, Weiss L, Bruel T, Zucman D, Appay V, Moris A, Ungeheuer MN, Lascoux-Combe C, Barre-Sinoussi F, Muller-Trutwin M, Boufassa F, Lambotte O, Pancino G, Saez-Cirion A; ANRS CO21 CODEX cohort. Dendritic Cells from HIV Controllers Have Low Susceptibility to HIV-1 Infection In Vitro but High Capacity to Capture HIV-1 Particles. PLoS One. 2016 Aug 9;11(8):e0160251. doi: 10.1371/journal.pone.0160251. eCollection 2016. PMID 27505169
- [Background] Duffy D, Rouilly V, Braudeau C, Corbiere V, Djebali R, Ungeheuer MN, Josien R, LaBrie ST, Lantz O, Louis D, Martinez-Caceres E, Mascart F, Ruiz de Morales JG, Ottone C, Redjah L, Guen NS, Savenay A, Schmolz M, Toubert A, Albert ML; Multinational FOCIS Centers of Excellence. Standardized whole blood stimulation improves immunomonitoring of induced immune responses in multi-center study. Clin Immunol. 2017 Oct;183:325-335. doi: 10.1016/j.clim.2017.09.019. Epub 2017 Sep 22. PMID 28943400
- [Background] Piasecka B, Duffy D, Urrutia A, Quach H, Patin E, Posseme C, Bergstedt J, Charbit B, Rouilly V, MacPherson CR, Hasan M, Albaud B, Gentien D, Fellay J, Albert ML, Quintana-Murci L; Milieu Interieur Consortium. Distinctive roles of age, sex, and genetics in shaping transcriptional variation of human immune responses to microbial challenges. Proc Natl Acad Sci U S A. 2018 Jan 16;115(3):E488-E497. doi: 10.1073/pnas.1714765115. Epub 2017 Dec 27. PMID 29282317
- [Background] Patin E, Hasan M, Bergstedt J, Rouilly V, Libri V, Urrutia A, Alanio C, Scepanovic P, Hammer C, Jonsson F, Beitz B, Quach H, Lim YW, Hunkapiller J, Zepeda M, Green C, Piasecka B, Leloup C, Rogge L, Huetz F, Peguillet I, Lantz O, Fontes M, Di Santo JP, Thomas S, Fellay J, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Publisher Correction: Natural variation in the parameters of innate immune cells is preferentially driven by genetic factors. Nat Immunol. 2018 Jun;19(6):645. doi: 10.1038/s41590-018-0105-3. PMID 29725081
- [Background] Scepanovic P, Alanio C, Hammer C, Hodel F, Bergstedt J, Patin E, Thorball CW, Chaturvedi N, Charbit B, Abel L, Quintana-Murci L, Duffy D, Albert ML, Fellay J; Milieu Interieur Consortium. Human genetic variants and age are the strongest predictors of humoral immune responses to common pathogens and vaccines. Genome Med. 2018 Jul 27;10(1):59. doi: 10.1186/s13073-018-0568-8. PMID 30053915
- [Background] Kilens S, Meistermann D, Moreno D, Chariau C, Gaignerie A, Reignier A, Lelievre Y, Casanova M, Vallot C, Nedellec S, Flippe L, Firmin J, Song J, Charpentier E, Lammers J, Donnart A, Marec N, Deb W, Bihouee A, Le Caignec C, Pecqueur C, Redon R, Barriere P, Bourdon J, Pasque V, Soumillon M, Mikkelsen TS, Rougeulle C, Freour T, David L; Milieu Interieur Consortium. Parallel derivation of isogenic human primed and naive induced pluripotent stem cells. Nat Commun. 2018 Jan 24;9(1):360. doi: 10.1038/s41467-017-02107-w. PMID 29367672
- [Background] Belizna C, Stojanovich L, Cohen-Tervaert JW, Fassot C, Henrion D, Loufrani L, Nagy G, Muchardt C, Hasan M, Ungeheuer MN, Arnaud L, Alijotas-Reig J, Esteve-Valverde E, Nicoletti F, Saulnier P, Godon A, Reynier P, Chretien JM, Damian L, Omarjee L, Mahe G, Pistorius MA, Meroni PL, Devreese K. Primary antiphospholipid syndrome and antiphospholipid syndrome associated to systemic lupus: Are they different entities? Autoimmun Rev. 2018 Aug;17(8):739-745. doi: 10.1016/j.autrev.2018.01.027. Epub 2018 Jun 6. PMID 29885541
- [Background] Belizna C, Pregnolato F, Abad S, Alijotas-Reig J, Amital H, Amoura Z, Andreoli L, Andres E, Aouba A, Apras Bilgen S, Arnaud L, Bienvenu B, Bitsadze V, Blanco P, Blank M, Borghi MO, Caligaro A, Candrea E, Canti V, Chiche L, Chretien JM, Cohen Tervaert JW, Damian L, Delross T, Dernis E, Devreese K, Djokovic A, Esteve-Valverde E, Favaro M, Fassot C, Ferrer-Oliveras R, Godon A, Hamidou M, Hasan M, Henrion D, Imbert B, Jeandel PY, Jeannin P, Jego P, Jourde-Chiche N, Khizroeva J, Lambotte O, Landron C, Latino JO, Lazaro E, de Leeuw K, Le Gallou T, Kilic L, Limper M, Loufrani L, Lubin R, Magy-Bertrand N, Mahe G, Makatsariya A, Martin T, Muchardt C, Nagy G, Omarjee L, Van Paasen P, Pernod G, Perrinet F, Pires Rosa G, Pistorius MA, Ruffatti A, Said F, Saulnier P, Sene D, Sentilhes L, Shovman O, Sibilia J, Sinescu C, Stanisavljevic N, Stojanovich L, Tam LS, Tincani A, Tollis F, Udry S, Ungeheuer MN, Versini M, Cervera R, Meroni PL. HIBISCUS: Hydroxychloroquine for the secondary prevention of thrombotic and obstetrical events in primary antiphospholipid syndrome. Autoimmun Rev. 2018 Dec;17(12):1153-1168. doi: 10.1016/j.autrev.2018.05.012. Epub 2018 Oct 12. PMID 30316994
- [Background] Prigent J, Lorin V, Kok A, Hieu T, Bourgeau S, Mouquet H. Scarcity of autoreactive human blood IgA+ memory B cells. Eur J Immunol. 2016 Oct;46(10):2340-2351. doi: 10.1002/eji.201646446. Epub 2016 Aug 25. PMID 27469325
- [Background] Bouchet J, Del Rio-Iniguez I, Vazquez-Chavez E, Lasserre R, Aguera-Gonzalez S, Cuche C, McCaffrey MW, Di Bartolo V, Alcover A. Rab11-FIP3 Regulation of Lck Endosomal Traffic Controls TCR Signal Transduction. J Immunol. 2017 Apr 1;198(7):2967-2978. doi: 10.4049/jimmunol.1600671. Epub 2017 Feb 24. PMID 28235866
- [Background] Aguera-Gonzalez S, Burton OT, Vazquez-Chavez E, Cuche C, Herit F, Bouchet J, Lasserre R, Del Rio-Iniguez I, Di Bartolo V, Alcover A. Adenomatous Polyposis Coli Defines Treg Differentiation and Anti-inflammatory Function through Microtubule-Mediated NFAT Localization. Cell Rep. 2017 Oct 3;21(1):181-194. doi: 10.1016/j.celrep.2017.09.020. PMID 28978472